CLINICAL TRIAL: NCT04992767
Title: Online Intervention to Promote Resilience to Traumatic Stress During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Jennifer Duffecy, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0002
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Posttraumatic Stress Disorder; Pregnancy Related
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sunnyside (Active Comparator): An online intervention to better manage mood during and after pregnancy.
  Interventions: Behavioral: Sunnyside
- SunnysideFlex (Experimental): An online intervention to treat symptoms of PTSD and better manage mood during and after pregnancy.
  Interventions: Behavioral: SunnysideFlex
- Treatment as Usual (No Intervention): A control condition consisting of standard prenatal medical care, without provision of the SunnysideFlex or Sunnyside intervention

INTERVENTIONS:
Behavioral: Sunnyside — The Sunnyside intervention is an online intervention(an interactive website with didactic material and interactive tools) targeting skills to manage mood during and after pregnancy. The Sunnyside intervention will consist of 6 weeks of online lessons during pregnancy and booster sessions at 2 weeks, 4 weeks, and 6 weeks postpartum. Each lesson takes approximately 10 minutes to complete.
  Arms: Sunnyside
Behavioral: SunnysideFlex — SunnysideFlex consists of 6 weeks of online lessons during pregnancy and booster sessions at 2 weeks, 4 weeks, and 6 weeks postpartum. SunnysideFlex has adapted the original Sunnyside intervention with revised, trauma-focused content that covers the impact of PTSD symptoms on the perinatal period and daily functioning, more broadly
  Arms: SunnysideFlex

SUMMARY:
The investigators will design, construct, and pilot a prototype of a trauma-informed online intervention, which will be called "SunnysideFlex," that functionally integrates a web-based intervention targeting skills to decrease symptoms of PTSD and better manage mood during and after pregnancy. SunnysideFlex will build upon the previously IRB-approved "Sunnyside" intervention which targeted skills to manage mood through an interactive website with didactic material and tools. Women in weeks 16-28 of their pregnancy who self-report symptoms of PTSD will be randomized to one of three study groups: (1) SunnysideFlex, (2) the original Sunnyside intervention (active control), or (3) treatment as usual (TAU). The SunnysideFlex intervention will consist of 6 weeks of trauma-informed online lessons during pregnancy and booster sessions at 2 weeks, 4 weeks, and 6 weeks postpartum. Outcomes will be measured at baseline, post-intervention, 6 weeks postpartum, and 12 weeks postpartum. SunnysideFlex has the potential to provide a novel paradigm for improving maternal and child health outcomes in high-risk, trauma-exposed women.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years and older
* Pregnant and between 16-28 weeks gestation
* Are currently engaged in prenatal care with a healthcare provider (OB/GYN, nurse, midwife, etc.)
* Endorse a history of one or more potentially traumatic events meeting Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) Criterion A for PTSD (i.e., "exposure to actual or threatened death, serious injury, or sexual violence," American Psychological Association [APA], p. 271) that is interpersonal in nature (e.g., sexual or physical assault, child abuse/maltreatment, witnessing family violence)
* Endorse a score of 33 or greater on the PTSD Checklist for DSM-5 (PCL-5)
* Have access to a broadband internet connection
* Able to read and speak English

Exclusion Criteria:

* Pregnant with multiples
* Have visual, hearing, voice, or motor impairment that would prevent completion of study procedures
* Have been diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, substance use disorder, or other diagnosis for which participation in this trial is either inappropriate or dangerous based on self-report
* Report currently being in an abusive or unsafe relationship
* Currently receiving treatment (medication or psychotherapy), or have an intention to resume antidepressant medication after delivery (i.e., women who discontinued their medication during pregnancy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Past 30 days
  The PCL-5 is a well validated screening tool for assessing PTSD symptoms and probable PTSD diagnosis. the PCL-5 checklist assesses frequency of past 30-day PTSD symptoms in reference to an individual's self-identified worst traumatic event. A total score of 33 or greater represents a positive PTSD screen and is the cut-off employed in the current study.
Impact of Events Scale - Revised (IES-R) | 1 week
  The IES-R assesses the past-week frequency of PTSD symptoms in reference to the participant's self-identified worst traumatic event
Patient Health Questionnaire-9 (PHQ-9) | 2 weeks
  Reflects overall functioning and impairment due to the depressive symptoms. PHQ-9 scoring interpretations are as follows: 1-4: minimal depressive symptoms; 5-9 mild depressive symptoms; 10-14: moderate depressive symptoms; 15-19: moderately severe depressive symptoms: 20-27: severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Duffecy, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Department of Psychology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No